CLINICAL TRIAL: NCT00005125
Title: NAS-NRC Twin Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 904
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2001-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Ischemia; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Ischemia; Obesity

SUMMARY:
To continue a registry of World War II veteran twins maintained by the National Academy of Sciences-National Research Council (NAS-NRC).

DETAILED DESCRIPTION:
BACKGROUND:

The registry of World War II veteran twins came into existence in the late 1960's through a search and link effort of state vital statistics records and Veterans Administration files through the Medical Follow-up Agency of NAS-NRC. Since that time, the registry has served as a data resource for investigators in a variety of scientific fields who want to study genetic and environmental aspects of various human characteristics. Because of the size and geographic coverage throughout the United States, the registry offers a method of recruiting sizeable numbers of twins for study even under geographic restrictions. Of special value to medical researchers is the built-in medical follow-up for morbidity and mortality through Veterans Administration insurance and benefits records. This allows researchers to gather baseline data which may be related prospectively to morbidity and mortality events.

The NHLBI has made extensive use of the World War II veteran twin registry beginning in 1969, when the NHLBI Twin Study was initiated. At that time, NHLBI used the World War II veteran twin registry to recruit a group of 514 pairs of twins in five geographic areas to participate in a study which included a battery of questionnaires and a physical examination. Since that time, a second examination and third examination of the cohort have been completed and the registry has been used to maintain contact with the twins and provide surveillance for morbidity and mortality events of the participants in the study.

DESIGN NARRATIVE:

Maintenance of the existing registry continued as addresses of all members were updated annually as well as morbidity and mortality data through surveillance of Veterans Administration insurance and death benefit records or through the National Death Index. All morbid events and deaths were coded by ICD codes. Support activities were provided for the NHLBI Twin Study including providing death certificates for events occurring among the 1,028 twins participating in the study and mailed questionnaire follow-up.

Although contract support ended in September, 1988, analyses of the survey and mortality data are continuing.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1970-07; Study Completion 1988-09

CONTACTS AND LOCATIONS:
Overall Officials: Zdenek Hrubec; Dennis Robinette

REFERENCES:
- [Background] Jablon S, Neel JV, Gershowitz H, Atkinson GF. The NAS-NRC twin panel: methods of construction of the panel, zygosity diagnosis, and proposed use. Am J Hum Genet. 1967 Mar;19(2):133-61. No abstract available. PMID 6067093
- [Background] Cederlof R, Friberg L, Hrubec Z. Cardiovascular and respiratory symptoms in relation to tobacco smoking. A study on American twins. Arch Environ Health. 1969 Jun;18(6):934-40. doi: 10.1080/00039896.1969.10665517. No abstract available. PMID 5770694
- [Background] Pollin W, Allen MG, Hoffer A, Stabenau JR, Hrubec Z. Psychopathology in 15,909 pairs of veteran twins: evidence for a genetic factor in the pathogenesis of schizophrenia and its relative absence in psychoneurosis. Am J Psychiatry. 1969 Nov;126(5):597-610. doi: 10.1176/ajp.126.5.597. No abstract available. PMID 5352613
- [Background] Allen MG, Pollin W. Schizophrenia in twins and the diffuse ego boundary hypothesis. Am J Psychiatry. 1970 Oct;127(4):437-42. doi: 10.1176/ajp.127.4.437. No abstract available. PMID 5459506
- [Background] Feinleib M, Havlik RJ, Kwiterovich PO, Tillotson J, Garrison RJ. The National Heart Institute Twin Study. Acta Genet Med Gemellol (Roma). 1970 Jan-Apr;19(1):243-7. doi: 10.1017/s1120962300025592. No abstract available. PMID 5533774
- [Background] Hoeffer A, Pollin W. Schizophrenia in the NAS-NRC panel of 15,909 veteran twin pairs. Arch Gen Psychiatry. 1970 Nov;23(5):469-77. doi: 10.1001/archpsyc.1970.01750050085012. No abstract available. PMID 5478575
- [Background] Reuling FH, Schwartz JT. Heritability of the effect of corticosteroids on intraocular pressure. Acta Genet Med Gemellol (Roma). 1970 Jan-Apr;19(1):264-7. doi: 10.1017/s1120962300025658. No abstract available. PMID 5533775
- [Background] Stabenau JR, Pollin W, Allen MG. Twin studies in schizophrenia and neurosis. Semin Psychiatry. 1970 Feb;2(1):65-74. No abstract available. PMID 5535862
- [Background] Cederlof R, Epstein FH, Friberg, et al: Twin Registries in the Study of Chronic Disease. Report of an International Symposium in San Juan, Puerto Rico, 1-4 December 1969, Acta Med Scand Suppl. 523, 1971
- [Background] Allen MG, Cohen S, Pollin W. Schizophrenia in veteran twins: a diagnostic review. Am J Psychiatry. 1972 Feb;128(8):939-45. doi: 10.1176/ajp.128.8.939. No abstract available. PMID 4550731
- [Background] Cohen SM, Allen MG, Pollin W, Hrubec Z. Relationship of schizo-affective psychosis to manic depressive psychosis and shizophrenia. Findings in 15,909 veteran pairs. Arch Gen Psychiatry. 1972 Jun;26(6):539-46. doi: 10.1001/archpsyc.1972.01750240051008. No abstract available. PMID 4554807
- [Background] Hrubec Z, Sutton ES. Smoking and health. Lancet. 1972 Oct 28;2(7783):932. doi: 10.1016/s0140-6736(72)92580-9. No abstract available. PMID 4116641
- [Background] Schwartz JT, Reuling FH, Feinleib M, Garrison RJ, Collie DJ. Twin heritability study of the effect of corticosteroids on intraocular pressure. J Med Genet. 1972 Jun;9(2):137-43. doi: 10.1136/jmg.9.2.137. No abstract available. PMID 5065285
- [Background] Hrubec Z. The effect of diagnostic ascertainment in twins on the assessment of the genetic factor in disease etiology. Am J Hum Genet. 1973 Jan;25(1):15-28. No abstract available. PMID 4684503
- [Background] Coffee drinking and ischaemic heart-disease. Lancet. 1973 Mar 10;1(7802):548-9. No abstract available. PMID 4119977
- [Background] Hrubec Z, Cederlof R, Friberg L, Horton R, Ozolins G. Respiratory symptoms in twins: effects of residence-associated air pollution, tobacco and alcohol use, and other factors. Arch Environ Health. 1973 Sep;27(3):189-95. doi: 10.1080/00039896.1973.10666350. No abstract available. PMID 4722874
- [Background] Schwartz JT, Reuling FH Jr, Feinleib M, Garrison RJ, Collie DJ. Twin heritability study of the corticosteroid response. Trans Am Acad Ophthalmol Otolaryngol. 1973 Mar-Apr;77(2):OP126-36. No abstract available. PMID 4738131
- [Background] Schwartz JT, Reuling FH, Feinleib M, Garrison RJ, Collie DJ. Twin study on ocular pressure after topical dexamethasone. 1. Frequency distribution of pressure response. Am J Ophthalmol. 1973 Jul;76(1):126-36. doi: 10.1016/0002-9394(73)90018-4. No abstract available. PMID 4736844
- [Background] Schwartz JT, Reuling FH, Feinleib M, Garrison RJ, Collie DJ. Twin study on ocular pressure following topically applied dexamethasone. II. Inheritance of variation in pressure response. Arch Ophthalmol. 1973 Oct;90(4):281-6. doi: 10.1001/archopht.1973.01000050283006. No abstract available. PMID 4795755
- [Background] Bazaral M, Orgel HA, and Hamburger RN: Genetics of IgE and Allergy: Serum IgE Levels in Twins. J Allergy Clin Immunol 54:288-304, 1974
- [Background] Lynfield YL. Skin diseases in twins. Arch Dermatol. 1974 Nov;110(5):722-4. No abstract available. PMID 4278385
- [Background] Bohning DE, Albert RE, Lippmann M, Foster WM. Tracheobronchial particle deposition and clearance. A study of the effects of cigarette smoking in monozygotic twins. Arch Environ Health. 1975 Sep;30(9):457-62. doi: 10.1080/00039896.1975.10666750. PMID 1172413
- [Background] Feinleib M, Garrison R, Borhani N, et al: Studies of Hypertension in Twins. In: Paul, Oglesby (Ed.): Epidemiology and Control of Hypertension, Second International Symposium on the Epidemiology of Hypertension, September 1974, Miami, Symposia Specialists, 1975
- [Background] Hrubec Z, Allen G. Letter: Methods and interpretation of twin concordance data. Am J Hum Genet. 1975 Nov;27(6):808-9. No abstract available. PMID 1239193
- [Background] Ziegler DK, Hassanein RS, Harris D, Stewart R. Headache in a non-clinic twin population. Headache. 1975 Jan;14(4):213-8. doi: 10.1111/j.1526-4610.1975.hed1404213.x. No abstract available. PMID 1123304
- [Background] Borhani NO, Feinleib M, Garrison RJ, Christian JC, Rosenman RH. Genetic variance in blood pressure. Acta Genet Med Gemellol (Roma). 1976;25:137-44. doi: 10.1017/s0001566000014008. PMID 1036353
- [Background] Christian JC, Feinleib M, Hulley SB, Castelli WP, Fabsitz RR, Garrison RJ, Borhani NO, Rosenman RH, Wagner J. Genetics of plasma cholesterol and triglycerides: a study of adult male twins. Acta Genet Med Gemellol (Roma). 1976;25:145-9. doi: 10.1017/s000156600001401x. PMID 1036354
- [Background] Feinleib M, Christian JC, Borhani NO, Rosenman R, Garrison RJ, Wagner J, Kannel WB, Hrubec Z, Schwartz JT. The National Heart and Lung Institute twin study of cardiovascular disease risk factors: organization and methodology. Acta Genet Med Gemellol (Roma). 1976;25:125-8. doi: 10.1017/s0001566000013970. No abstract available. PMID 1036351
- [Background] Horn JM, Plomin R, Rosenman R. Heritability of personality traits in adult male twins. Behav Genet. 1976 Jan;6(1):17-30. doi: 10.1007/BF01065675. PMID 943159
- [Background] Hrubec Z, Cederlof R, Friberg L. Background of angina pectoris: social and environmental factors in relation to smoking. Am J Epidemiol. 1976 Jan;103(1):16-29. doi: 10.1093/oxfordjournals.aje.a112201. PMID 1247009
- [Background] Rosenman RH, Rahe RH, Borhani NO, Feinleib M. Heritability of personality and behavior pattern. Acta Genet Med Gemellol (Roma). 1976;25:221-4. doi: 10.1017/s0001566000014161. PMID 1036367
- [Background] Taubman P: The Determinants of Earnings: Genetics, Family and Other Environments. A Study of White Male Twins. Am Economic Rev 66:858-870, 1976
- [Background] Taubman P. Earnings, education, genetics, and environment. J Hum Resour. 1976 Fall;11(4):447-61. PMID 988067
- [Background] Behrman J, Taubman P, and Wales T: Controlling For and Measuring the Effects of Genetics and Family Environment in Equations for Schooling and Labor Market Success. In: Taubman P (Ed.): Kinometrics: Determinants of Socioeconomic Success Within and Between Families, New York, North-Holland Publishing Company, 1977
- [Background] Feinleib M, Garrison RJ, Fabsitz R, Christian JC, Hrubec Z, Borhani NO, Kannel WB, Rosenman R, Schwartz JT, Wagner JO. The NHLBI twin study of cardiovascular disease risk factors: methodology and summary of results. Am J Epidemiol. 1977 Oct;106(4):284-5. doi: 10.1093/oxfordjournals.aje.a112464. PMID 562066
- [Background] Havlik R, Garrison R, Fabsitz R, Feinleib M. Genetic variability of clinical chemical values. Clin Chem. 1977;23(4):659-62. PMID 557378
- [Background] Bobowick AR, Kurtzke JF, Brody JA, Hrubec Z, Gillespie M. Twin study of multiple sclerosis: an epidemiologic inquiry. Neurology. 1978 Oct;28(10):978-87. doi: 10.1212/wnl.28.10.978. PMID 570667
- [Background] Fabsitz RR, Garrison RJ, Feinleib M, Hjortland M. A twin analysis of dietary intake: evidence for a need to control for possible environmental differences in MZ and DZ twins. Behav Genet. 1978 Jan;8(1):15-25. doi: 10.1007/BF01067701. PMID 565201
- [Background] Feinleib M, Ware JH, Garrison RJ, Borhani N, Christian JC, Rosenman R. An analysis of variance for major coronary heart disease rick factors in twins and their brothers. Prog Clin Biol Res. 1978;24 Pt C:13-9. No abstract available. PMID 569315
- [Background] Hrubec Z, Neel JV. The National Academy of Sciences--National Research Council Twin Registry: ten years of operation. Prog Clin Biol Res. 1978;24 Pt B:153-72. No abstract available. PMID 569304
- [Background] Rahe RH, Hervig L, Rosenman RH. Heritability of type A behavior. Psychosom Med. 1978 Oct;40(6):478-86. doi: 10.1097/00006842-197810000-00003. PMID 569878
- [Background] Taubman P: What We Learn from Estimating the Genetic Contribution to Inequality in Earnings: Reply, Am Econ Rev 68:970-976, 1978
- [Background] Allen G, Hrubec Z. Twin concordance. A more general model. Acta Genet Med Gemellol (Roma). 1979;28(1):3-13. doi: 10.1017/s0001566000009284. PMID 575693
- [Background] Anderson RE, Hill RB, and Hrubec Z: Prospects for Pathology Studies in the NAS-NRC Twin Registry. Hum Pathol 11:403, 1980
- [Background] Fabsitz R, Feinleib M, Hrubec Z. Weight changes in adult twins. Acta Genet Med Gemellol (Roma). 1980;29(4):273-9. doi: 10.1017/s0001566000007789. PMID 7197452
- [Background] Foch TT, and McClearn GE: Genetics, Body Weight, and Obesity. In: Stunkard, AJ (Ed.): Obesity, Philadelphia, Saunders Publishing Company, pp. 48-71, 1980
- [Background] Havlik RJ, Garrison RJ, Fabsitz R, Feinleib M. Variability of heart rate, P-R, QRS and Q-T durations in twins. J Electrocardiol. 1980;13(1):45-8. doi: 10.1016/s0022-0736(80)80008-2. PMID 7188949
- [Background] Hrubec Z, and Omenn GS: Evidence of Genetic Predisposition to Alcoholic Cirrhosis and Psychosis: Twin Concordances for Alcoholism and Its Biologic End Points by Zygosity Among Male Veterans (Abstract of paper presented at Thirty-first Annual Meeting, American Society of Human Genetics, New York, September 1980), Am J Hum Genet 32:112A, 1980
- [Background] Hubert HB, Fabsitz RR, Feinleib M, Brown KS. Olfactory sensitivity in humans: genetic versus environmental control. Science. 1980 May 9;208(4444):607-9. doi: 10.1126/science.7189296.
- [Background] Hrubec Z: Methodologic Problems in Matched-Pair Studies Using Twins. In: Gedda L, Parisi P, and Nance WE (Eds.): Twin Research 3. Proceedings of the Third International Congress on Twin Studies, June 16-20, 1980, Jerusalem, Part C. Epidemiological and Clinical Studies, Progress in Clinical and Biological Research Volume 69C, New York, Alan R. Liss, Inc., pp. 1-7, 1981
- [Background] Hrubec Z, Neel JV. Familial factors in early deaths: twins followed 30 years to ages 51-61 in 1978. Hum Genet. 1981;59(1):39-46. doi: 10.1007/BF00278852. PMID 10819020
- [Background] Hrubec Z, Omenn GS. Evidence of genetic predisposition to alcoholic cirrhosis and psychosis: twin concordances for alcoholism and its biological end points by zygosity among male veterans. Alcohol Clin Exp Res. 1981 Spring;5(2):207-15. doi: 10.1111/j.1530-0277.1981.tb04890.x. PMID 7018299
- [Background] Hrubec Z, Neel JV. Contribution of familial factors to the occurrence of cancer before old age in twin veterans. Am J Hum Genet. 1982 Jul;34(4):658-71. PMID 7201741
- [Background] Kendler KS, Robinette CD. Schizophrenia in the National Academy of Sciences-National Research Council Twin Registry: a 16-year update. Am J Psychiatry. 1983 Dec;140(12):1551-63. doi: 10.1176/ajp.140.12.1551. PMID 6685980
- [Background] Kendler KS, Robinette CD. Month of birth by zygosity in the NAS-NRC twin registry. Acta Genet Med Gemellol (Roma). 1983;32(2):113-6. doi: 10.1017/s0001566000006395. PMID 6650099
- [Background] Fabsitz R, Feinleib M, Hubert H. Regression analysis of data with correlated errors: an example from the NHLBI twin study. J Chronic Dis. 1985;38(2):165-70. doi: 10.1016/0021-9681(85)90089-x. PMID 4038711
- [Background] Matthews KA, Rosenman RH, Dembroski TM, Harris EL, MacDougall JM. Familial resemblance in components of the type A behavior pattern: a reanalysis of the California type A twin study. Psychosom Med. 1984 Nov-Dec;46(6):512-22. doi: 10.1097/00006842-198411000-00004. PMID 6542684
- [Background] Hrubec Z, Robinette CD. The study of human twins in medical research. N Engl J Med. 1984 Feb 16;310(7):435-41. doi: 10.1056/NEJM198402163100706. No abstract available. PMID 6363927
- [Background] Carmelli D, Chesney MA, Ward MM, Rosenman RH. Twin similarity in cardiovascular stress response. Health Psychol. 1985;4(5):413-23. doi: 10.1037//0278-6133.4.5.413. PMID 4076117
- [Background] Kalousdian S, Fabsitz R, Havlik R, Christian J, Rosenman R. Heritability of clinical chemistries in an older twin cohort: the NHLBI Twin Study. Genet Epidemiol. 1987;4(1):1-11. doi: 10.1002/gepi.1370040102. PMID 3569874
- [Background] Luxenberg JS, May C, Haxby JV, Grady C, Moore A, Berg G, White BJ, Robinette D, Rapoport SI. Cerebral metabolism, anatomy, and cognition in monozygotic twins discordant for dementia of the Alzheimer type. J Neurol Neurosurg Psychiatry. 1987 Mar;50(3):333-40. doi: 10.1136/jnnp.50.3.333. PMID 3494105
- [Background] Carmelli D, Rosenman R, Chesney M, Fabsitz R, Lee M, Borhani N. Genetic heritability and shared environmental influences of type A measures in the NHLBI Twin Study. Am J Epidemiol. 1988 May;127(5):1041-52. doi: 10.1093/oxfordjournals.aje.a114880. PMID 3358405
- [Background] Selby JV, Newman B, Quesenberry CP Jr, Fabsitz RR, King MC, Meaney FJ. Evidence of genetic influence on central body fat in middle-aged twins. Hum Biol. 1989 Apr;61(2):179-94. PMID 2767669
- [Background] Christian JC, Carmelli D, Castelli WP, Fabsitz R, Grim CE, Meaney FJ, Norton JA Jr, Reed T, Williams CJ, Wood PD. High density lipoprotein cholesterol. A 16-year longitudinal study in aging male twins. Arteriosclerosis. 1990 Nov-Dec;10(6):1020-5. doi: 10.1161/01.atv.10.6.1020. PMID 2244851
- [Background] Selby JV, Newman B, Quesenberry CP Jr, Fabsitz RR, Carmelli D, Meaney FJ, Slemenda C. Genetic and behavioral influences on body fat distribution. Int J Obes. 1990 Jul;14(7):593-602. PMID 2228394
- [Background] Carmelli D, Swan GE, Robinette D, Fabsitz RR. Heritability of substance use in the NAS-NRC Twin Registry. Acta Genet Med Gemellol (Roma). 1990;39(1):91-8. doi: 10.1017/s0001566000005602. PMID 2392895
- [Background] Swan GE, Carmelli D, Reed T, Harshfield GA, Fabsitz RR, Eslinger PJ. Heritability of cognitive performance in aging twins. The National Heart, Lung, and Blood Institute Twin Study. Arch Neurol. 1990 Mar;47(3):259-62. doi: 10.1001/archneur.1990.00530030025010. PMID 2310310
- [Background] Reed T, Fabsitz RR, Quiroga J. Family history of ischemic heart disease with respect to mean twin-pair cholesterol and subsequent ischemic heart disease in the NHLBI twin study. Genet Epidemiol. 1990;7(5):335-47. doi: 10.1002/gepi.1370070504. PMID 2253868
- [Background] Newman B, Selby JV, Quesenberry CP Jr, King MC, Friedman GD, Fabsitz RR. Nongenetic influences of obesity on other cardiovascular disease risk factors: an analysis of identical twins. Am J Public Health. 1990 Jun;80(6):675-8. doi: 10.2105/ajph.80.6.675. PMID 2343948
- [Background] Havlik RJ, Fabsitz RR, Kalousdian S, Borhani NO, Christian JC. Dietary protein and blood pressure in monozygotic twins. Prev Med. 1990 Jan;19(1):31-9. doi: 10.1016/0091-7435(90)90004-4. PMID 2320557
- [Background] DeCarli C, Miller BL, Swan GE, Reed T, Wolf PA, Carmelli D. Cerebrovascular and brain morphologic correlates of mild cognitive impairment in the National Heart, Lung, and Blood Institute Twin Study. Arch Neurol. 2001 Apr;58(4):643-7. doi: 10.1001/archneur.58.4.643. PMID 11295996